CLINICAL TRIAL: NCT02437383
Title: Effect of COMT (Catecholamine-O-methyltransferase) Genetic Polymorphisms on Response to Propranolol Therapy in Temporomandibular Disorder
Brief Title: Study of Orofacial Pain and PropRANOlol
Acronym: SOPPRANO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: University of Florida (Other); Rho, Inc. (Industry); National Institutes of Health (NIH) (NIH); National Institute of Dental and Craniofacial Research (NIDCR) (NIH); State University of New York at Buffalo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 14-2526; 1U01DE024169-01 (NIH); 14-067-E (Other: NIDCR Protocol Number)
Record Dates: First submitted 2015-05-04; First posted 2015-05-07 (Estimated); Results first posted 2019-05-21 (Actual); Last update posted 2019-05-21 (Actual); Status verified 2018-04

CONDITIONS: Temporomandibular Disorders
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Propranolol; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Propranolol ER (Active Comparator): Propranolol hydrochloride extended release (ER) capsules; 60 mg (Visit 1 and Visit 4); 120 mg (Visit 2 and Visit 3) given orally as: 60 mg once/day (Visit 1 and Visit 4) and 60 mg twice/day (Visit 2 and Visit 3).
  Interventions: Drug: Propranolol ER
- Placebo (Placebo Comparator): Capsules, identical in appearance to active comparator (propranolol), to be administered orally in exactly the same manner as propranolol at Visit 1 (once/day), Visit 2 (twice/day), Visit 3 (twice/day), and Visit 4 (once/day).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Propranolol ER — Capsules given orally according to schedule at Visit 1, Visit 2, Visit 3, and Visit 4.
  Other Names: Inderal (long-acting)
  Arms: Propranolol ER
Drug: Placebo — Gelatin capsules with a microcrystalline cellulose filler manufactured to mimic propranolol ER 60 mg capsules
  Other Names: Sugar pill
  Arms: Placebo

SUMMARY:
Purpose:

Primary: To evaluate the efficacy of extended-release (ER) propranolol compared to placebo in the reduction of a pain index in patients with temporomandibular disorder (TMD).

Secondary: To determine if extended-release propranolol efficacy varies according to participants' catechol-O-methyltransferase (COMT) genetic polymorphisms and to investigate the efficacy of extended-release propranolol compared with placebo using secondary endpoints.

Exploratory: To investigate whether the efficacy of extended-release propranolol in the reduction of the pain index varies according to participants' polymorphisms in 3 other genetic regions and according to various phenotypic characteristics.

Participants:

200 patients with chronic TMD will be randomly assigned, in a 1:1 parallel, double-blind fashion, to receive either extended-release propranolol or placebo at one of three study sites: University of North Carolina-Chapel Hill School of Dentistry; University of Florida-Gainesville College of Dentistry; and the State University of New York at Buffalo School of Dental Medicine.

Procedures (methods):

Randomization will be to either propranolol or placebo. The 10-week study treatment period is divided into: 1 week of drug titration, 8 weeks of drug maintenance, and 1 week of drug tapering. The titration and tapering doses are 60 mg (capsules) once per day orally; the maintenance dose is 60 mg twice per day orally. Participants will attend 6 clinic visits over 12-15 weeks as follows: screening and baseline visit (Visit [V] 0, 7-21 days prior to V1); randomization and start of treatment (titration) (V1, study day 0); maintenance visit 2 (V2, 1 week post-randomization, study day 7+3); maintenance visit 3 (V3, 5 weeks post-randomization, study day 35 +/- 7); tapering visit (V4, 9 weeks post-randomization, study day 63 +/- 7); and tapering visit 5 (V5, 11 weeks post-randomization and 1 week after drug tapering ends, study day 77 +/- 7). Depending on the visit, procedures will include: reviews of medical history, weekly alcohol consumption, concomitant therapies and medications, adverse events, compliance, and eligibility; administration/review of questionnaires; blood draw; pregnancy test in women of childbearing potential; and dispensing of study drug.

DETAILED DESCRIPTION:
"Temporomandibular disorder" (TMD) encompasses all musculoskeletal disorders of the masticatory system and includes myalgia, arthralgia, temporomandibular joint (TMJ) disc displacements, and TMJ degenerative joint diseases. The prevalence of TMD ranges from 6% to 12% in the general population, with muscle dysfunction the most prevalent TMD diagnostic group. TMD is associated with substantial disability and suffering and negatively impacts quality of life. Jaw pain is the most common symptom that compels treatment seeking. In addition to facial pain, TMD patients frequently report comorbid pain conditions such as headache, low back pain, and fibromyalgia. New approaches to TMD therapy are urgently needed to improve clinical outcomes and reduce economic impact of this disorder.

There is currently no FDA-approved product labeled specifically to manage/treat TMD; however, classes of drugs are used to relieve TMD-associated pain, such as non-steroidal anti-inflammatory drugs (NSAIDs), anti-inflammatory drugs, corticosteroids, benzodiazepines, sedative hypnotics, muscle relaxants, opioids, antidepressants, and anticonvulsants - although evidence to establish their efficacy and safety in this population is scarce. Practitioners' justification for their use may be based on poorly controlled clinical trials or clinical trials in other pain disorders such as acute postsurgical dental pain, arthritic pain, chronic lower back pain, and neuropathic pain. Thus, there is a need for controlled clinical trials to better understand the physiological mechanisms responsible for TMD symptoms.

Evidence suggests that enhanced β-adrenergic drive contributes to the pathogenesis of TMD and other complex persistent pain conditions. For example, individuals with myofascial pain conditions have elevated catecholamine levels and augmented sympathetic responses to stressors. While increased β-adrenergic drive appears to heighten pain, β-adrenergic antagonists can reduce clinical pain and/or nociceptive sensitivity. A recent study of a single infusion of propranolol in TMD and fibromyalgia patients revealed short-term improvement in clinical pain ratings. The antagonist pindolol was similarly efficacious in alleviating cardinal symptoms of fibromyalgia pain. In addition, intramuscular injections of low-dose propranolol in rats reduced inflammatory pain associated with carrageen-induced inflammation of the gastrocnemius muscle.

The study hypothesis is that therapy with the nonselective β-adrenergic receptor antagonist propranolol extended-release capsules (FDA approved to treat many cardiac conditions, tremor, migraine, and pheochromocytoma) will provide efficacious and safe treatment for painful TMD. It has well-studied pharmacodynamic, pharmacokinetic, and side-effect profiles. Peak blood level occurs at approximately 6 hrs, and the plasma half-life is approximately 10 hrs. The primary objective is to investigate the efficacy of propranolol compared with placebo over 9 weeks to reduce pain in patients with TMD. Secondary objectives are to: investigate by treatment group whether reduction in pain varies according to polymorphisms in the COMT gene coding region; and investigate the effect of propranolol compared with placebo to affect pain sensitivity, physical and emotional function, adverse effects, and use of rescue medications. Exploratory objectives are to: investigate gene-by-treatment group interaction to determine the effect of propranolol on reduction in the pain index according to polymorphisms in the COMT, beta-2 adrenergic receptor (ADRβ2), and beta-3 adrenergic receptor (ADRβ3) genetic coding regions.

ELIGIBILITY:
Inclusion:

* Diagnostic criteria for TMD: Group II, Masticatory Muscle Disorders, Myalgia
* Facial pain for at least 3 months (and at least 10 of the last 30 days at Visit 0)
* Average pain intensity rating ≥30 (0-100 numeric rating scale) over the past week or average daily pain intensity rating ≥30 on the same scale on at least 3 days over the past week
* Agrees to terms for continuing/discontinuing certain prescription/over-the-counter pain medications throughout participation
* Agrees to not commence new prescription medication, injection therapy, occlusal splint therapy or certain other pain management techniques throughout participation
* Agrees to limit consumption of alcohol to no more than 7 drinks/week (females) and no more than 14 drinks/week (males) throughout participation
* If a female of childbearing potential, agrees to use of contraception (licensed hormonal method, intrauterine device, condoms with contraceptive foam, abstinence, or partner vasectomy) throughout participation
* Able to understand and comply with study procedures and provide written informed consent

Exclusion:

* History of congestive heart failure or certain cardiac conditions including coronary artery disease, uncontrolled hypertension, or hypotension
* Bronchial asthma, nonallergic bronchospasm, renal failure or dialysis, diabetes mellitus, hyperthyroidism, fibromyalgia, or uncontrolled seizures
* Currently taking a β-blocker or certain other medications including haloperidol, intravenous verapamil, or reserpine
* Currently taking an opioid medication
* Daily prescription medication, occlusal splint therapy, or an investigational drug or treatment for pain management within past 30 days
* Injection therapy or certain other pain management techniques within last 2 weeks
* Facial trauma or orofacial surgery within past 6 weeks
* Active orthodontic treatment
* History of major depression or other psychiatric disorder requiring hospitalization within past 6 months
* Treatment for drug or alcohol abuse within the last year
* Smokes 25 or more cigarettes/day
* Currently receiving chemotherapy or radiation therapy
* Pregnant or breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2015-08-20 (Actual); Primary Completion 2018-04-04 (Actual); Study Completion 2018-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Inna E. Tchivileva, MD, Principal Investigator — University of North Carolina, Chapel Hill; Roger B. Fillingim, PhD, Principal Investigator — University of Florida-Gainesville College of Dentistry; Richard Ohrbach, DDS, PhD, Principal Investigator — University at Buffalo School of Dental Medicine
Locations (3):
- United States (3):
  - University of Florida-Gainesville College of Dentistry, Gainesville, Florida
  - University at Buffalo School of Dental Medicine, Buffalo, New York
  - University of North Carolina at Chapel Hill School of Dentistry, Chapel Hill, North Carolina

REFERENCES:
- [Background] Tchivileva IE, Lim PF, Smith SB, Slade GD, Diatchenko L, McLean SA, Maixner W. Effect of catechol-O-methyltransferase polymorphism on response to propranolol therapy in chronic musculoskeletal pain: a randomized, double-blind, placebo-controlled, crossover pilot study. Pharmacogenet Genomics. 2010 Apr;20(4):239-48. doi: 10.1097/FPC.0b013e328337f9ab. PMID 20216107
- [Background] Gursoy S, Erdal E, Herken H, Madenci E, Alasehirli B, Erdal N. Significance of catechol-O-methyltransferase gene polymorphism in fibromyalgia syndrome. Rheumatol Int. 2003 May;23(3):104-7. doi: 10.1007/s00296-002-0260-5. Epub 2002 Oct 22. PMID 12739038
- [Background] Diatchenko L, Slade GD, Nackley AG, Bhalang K, Sigurdsson A, Belfer I, Goldman D, Xu K, Shabalina SA, Shagin D, Max MB, Makarov SS, Maixner W. Genetic basis for individual variations in pain perception and the development of a chronic pain condition. Hum Mol Genet. 2005 Jan 1;14(1):135-43. doi: 10.1093/hmg/ddi013. Epub 2004 Nov 10. PMID 15537663
- [Derived] Tchivileva IE, Ohrbach R, Fillingim RB, Lin FC, Lim PF, Arbes SJ Jr, Slade GD. Clinical, psychological, and sensory characteristics associated with headache attributed to temporomandibular disorder in people with chronic myogenous temporomandibular disorder and primary headaches. J Headache Pain. 2021 May 22;22(1):42. doi: 10.1186/s10194-021-01255-1. PMID 34022805
- [Derived] Tchivileva IE, Ohrbach R, Fillingim RB, Lim PF, Giosia MD, Ribeiro-Dasilva M, Campbell JH, Hadgraft H, Willis J, Arbes SJ Jr, Slade GD. Effect of comorbid migraine on propranolol efficacy for painful TMD in a randomized controlled trial. Cephalalgia. 2021 Jun;41(7):839-850. doi: 10.1177/0333102421989268. Epub 2021 Feb 9. PMID 33560875
- [Derived] Slade GD, Fillingim RB, Ohrbach R, Hadgraft H, Willis J, Arbes SJ Jr, Tchivileva IE. COMT Genotype and Efficacy of Propranolol for TMD Pain: A Randomized Trial. J Dent Res. 2021 Feb;100(2):163-170. doi: 10.1177/0022034520962733. Epub 2020 Oct 8. PMID 33030089
- [Derived] Tchivileva IE, Hadgraft H, Lim PF, Di Giosia M, Ribeiro-Dasilva M, Campbell JH, Willis J, James R, Herman-Giddens M, Fillingim RB, Ohrbach R, Arbes SJ Jr, Slade GD. Efficacy and safety of propranolol for treatment of temporomandibular disorder pain: a randomized, placebo-controlled clinical trial. Pain. 2020 Aug;161(8):1755-1767. doi: 10.1097/j.pain.0000000000001882. PMID 32701836
- [Derived] Sanders AE, Slade GD, Fillingim RB, Ohrbach R, Arbes SJ Jr, Tchivileva IE. Effect of Treatment Expectation on Placebo Response and Analgesic Efficacy: A Secondary Aim in a Randomized Clinical Trial. JAMA Netw Open. 2020 Apr 1;3(4):e202907. doi: 10.1001/jamanetworkopen.2020.2907. PMID 32297945

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Propranolol ER | Placebo
Started | 100 | 100
Completed | 87 | 87
Not Completed | 13 | 13

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of treatment and provided at least one post-baseline data point (N=199). No data were available for one randomized participant in the placebo arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | Propranolol ER | Placebo | Total
Number analyzed (Participants) | 100 | 99 | 199
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.9 (12.19) | 34.2 (13.29) | 34.1 (12.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 78 | 155
  Male | 23 | 21 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 8 | 12
  Not Hispanic or Latino | 93 | 89 | 182
  Unknown or Not Reported | 3 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 6 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Black or African American | 12 | 18 | 30
  White | 79 | 71 | 150
  More than one race | 2 | 2 | 4
  Unknown or Not Reported | 2 | 0 | 2
Weekly Mean Pain Intensity [Mean (Standard Deviation); unit: units on a scale] — Weekly mean pain intensity computed as the arithmetic mean of daily pain intensity values during the week prior to randomization. Daily pain intensity is measured on 0-100 numeric rating scale where 0 = "no pain" and 100 = "the most intense pain imaginable") as reported in the Daily Symptom Diary. A higher score means a worse outcome.
  units on a scale | 47.9 (15.23) | 47.4 (15.58) | 47.6 (15.37)
Weekly Mean Pain Duration [Mean (Standard Deviation); unit: units on a scale] — Weekly mean pain duration computed as the arithmetic mean of daily pain duration values during the week prior to randomization. Daily pain duration is measured on 0-100 percentage scale where percent = "percent of waking day you had facial pain" as reported in the Daily Symptom Diary. A higher score means a worse outcome.
  units on a scale | 56.6 (26.57) | 60.1 (24.61) | 58.3 (25.61)
Weekly Mean Pain Index [Mean (Standard Deviation); unit: units on a scale] — Weekly mean pain index computed as the arithmetic mean of daily pain index values during the week prior to randomization. Daily pain index is computed as pain intensity (0-100 numeric rating scale where 0 = "no pain" and 100 = "the most intense pain imaginable") multiplied by pain duration (0-100 percentage scale where percent = "percent of waking day you had facial pain") as reported in the Daily Symptom Diary, divided by 100. The pain index range is from 0 to 100. A higher score means a worse outcome.
  units on a scale | 30.0 (19.96) | 31.2 (18.94) | 30.6 (19.42)
The SF-McGill Pain Questionnaire Affective Component [Mean (Standard Deviation); unit: units on a scale] — The SF-McGill Pain Questionnaire contains 4 affective descriptors rated on a 0-3 scale where 0 = "none," 1 = "mild," 2 = "moderate," and 3 = "severe."The item scores are summed to yield a total score with a range from 0 to 12. A higher score means a worse outcome.
  units on a scale | 3.5 (2.22) | 3.4 (2.33) | 3.4 (2.27)
The SF-McGill Pain Questionnaire Sensory Component [Mean (Standard Deviation); unit: units on a scale] — The SF-McGill Pain Questionnaire contains 11 sensory descriptors rated on a 0-3 scale where 0 = "none," 1 = "mild," 2 = "moderate," and 3 = "severe."The item scores are summed to yield a total score with a range form 0 to 33. A higher score means a worse outcome.
  units on a scale | 5.1 (6.40) | 4.8 (6.12) | 5.0 (6.25)
The SF-McGill Pain Questionnaire Present Facial Pain Intensity [Mean (Standard Deviation); unit: units on a scale] — Self-reported present intensity of facial pain at the moment of assessment scored on a descriptive scale where 1 = "no pain' and 6 = "excruciating pain." A higher score means worse outcome.
  units on a scale | 3.0 (0.87) | 3.0 (0.93) | 3.0 (0.90)
The SF-McGill Pain Questionnaire Weekly Average Facial Pain Intensity [Mean (Standard Deviation); unit: units on a scale] — Self-reported average facial pain intensity for the last week scored on 0-100 numerical rating scale where 0 = "no pain" and 100 = "the most intense pain imaginable". A higher score means a worse outcome.
  units on a scale | 56.0 (16.55) | 56.2 (17.41) | 56.1 (16.94)
The SF-McGill Pain Questionnaire Weekly Average Facial Pain Duration [Mean (Standard Deviation); unit: units on a scale] — Self-reported average facial pain duration for the last week scored on 0-100 percentage scale where percent = "percent of waking day you had facial pain." A higher score means a worse outcome.
  units on a scale | 63.2 (29.22) | 67.0 (23.93) | 65.1 (26.72)
The SF-McGill Pain Questionnaire Weekly Fatigue [Mean (Standard Deviation); unit: units on a scale] — Self-reported average fatigue for the last week scored on 0-100 numerical rating scale where 0 = "no fatigue" and 100 = "the greatest imaginable." A higher score means a worse outcome.
  units on a scale | 41.8 (26.75) | 41.1 (28.36) | 41.4 (27.49)
Number of Participants Stratified per Graded Chronic Pain Scale (GCPS) grade [Count of Participants; unit: Participants] — Individuals were classified into 6 chronic pain grades: 0 = no pain; I = low pain intensity and low pain-related disability; IIa = high pain intensity and low pain-related disability; IIb = high pain intensity and high activity interference; III = moderate pain-related disability; and IV = severe pain-related disability. For analyses, this variable was dichotomized: grades 0-IIa were combined in one category and all higher grades in another. A higher grade means a worse outcome.
  Participants
    GCPS Grades 0-IIa | 59 | 57 | 116
    GCPS Grades IIb-IV | 41 | 42 | 83
The Jaw Functional Limitation Scale (JFLS) Global Score [Mean (Standard Deviation); unit: units on a scale] — The JFLS contains 20 items that measure limitations across mastication, vertical jaw mobility, and verbal/emotional expression rated on a 0-10 scale where 0 = "no limitation" and 10 = "severe limitation." The Global Score is computed as the mean response for all items and ranges from 0 to 10. A higher score means a worse outcome.
  units on a scale | 2.8 (1.76) | 2.5 (1.52) | 2.6 (1.64)
The Headache Impact Test (HIT-6) Global Score [Mean (Standard Deviation); unit: units on a scale] — The HIT-6 contains 6 items and assesses headache-related disability by the frequency of daily activity limitations ranging from "never" to "always." The 6 item scores are summed to yield a global score ranging from 36 to 78. A higher score means a worse outcome.
  units on a scale | 54.4 (9.10) | 55.2 (8.70) | 54.8 (8.89)
The Perceived Stress Scale (PSS) Global Score [Mean (Standard Deviation); unit: units on a scale] — The PSS assesses the frequency of 14 sources of stress on a scale from 0 = "never" to 4 = "very often." The item scores are summed to yield a Global Score ranging from 0 to 56. A higher score means a worse outcome.
  units on a scale | 21.2 (8.99) | 21.5 (9.12) | 21.3 (9.03)
The Pittsburgh Sleep Quality Index (PSQI) Global Score [Mean (Standard Deviation); unit: units on a scale] — The PSQI has 19 items grouped into 7 component scores, each weighted equally on a 0-3 scale, The 7 component scores are summed to yield a global PSQI score, which has a range of 0-21. A higher score means a worse outcome.
  units on a scale | 6.5 (3.66) | 6.6 (3.58) | 6.5 (3.61)
The Hospital Anxiety and Depression Scale (HADS) Anxiety Score [Mean (Standard Deviation); unit: units on a scale] — The HADS is a 14-item assessment of anxiety (7 items) and depression (7 items) using the relative frequency of symptoms over the past week, rated on a 4-point scale ranging from 0 = "not at all" to 3 = "very often indeed". Responses are summed to provide separate scores for anxiety and depression (range from 0 to 21 for each subscale). A higher score means a worse outcome.
  units on a scale | 6.9 (4.19) | 7.5 (4.59) | 7.2 (4.39)
The Hospital Anxiety and Depression Scale (HADS) Depression Score [Mean (Standard Deviation); unit: units on a scale] — The HADS is a 14-item assessment of anxiety (7 items) and depression (7 items) using the relative frequency of symptoms over the past week, rated on a 4-point scale ranging from 0 = "not at all" to 3 = "very often indeed". Responses are summed to provide separate scores for anxiety and depression (range from 0 to 21 for each subscale). A higher score means a worse outcome.
  units on a scale | 3.7 (3.54) | 3.3 (3.14) | 3.5 (3.35)
The Symptom Checklist 90-Revised (SCL-90R) Somatization Scale Score [Mean (Standard Deviation); unit: units on a scale] — The SCL-90R Somatization Scale is a 12-item assessment of somatic symptom distress over the past 7 days rated from 0 = "not at all" to 4 = "extremely." The scale score is computed as the mean for all items. The score range is from 0 to 4. The higher score means a worse outcome.
  units on a scale | 0.6 (0.50) | 0.7 (0.51) | 0.6 (0.50)
The SF-12 Health Survey v2 (SF-12v2) Physical Component Summary (PCS) [Mean (Standard Deviation); unit: units on a scale] — The SF-12v2 v2 contains 7 questions assessing 8 domains of functioning and well-being rated from: "excellent" to "poor" (for general health); "yes, limited a lot" to "no, not limited at all" (for functional level); and "all of the time" to "none of the time" (for emotional state). These 8 domains can be further summarized into a physical component summary (PCS) and a mental component summary (MCS). The range for each component is 0-100 and a higher score means a better outcome.
  units on a scale | 48.4 (10.71) | 50.0 (9.39) | 49.2 (10.08)
The SF-12 Health Survey v2 (SF-12v2) Mental Component Summary (MCS) [Mean (Standard Deviation); unit: units on a scale] — The SF-12v2 v2 contains 7 questions assessing 8 domains of functioning and well-being rated from: "excellent" to "poor" (for general health); "yes, limited a lot" to "no, not limited at all" (for functional level); and "all of the time" to "none of the time" (for emotional state). These 8 domains can be further summarized into a physical component summary (PCS) and a mental component summary (MCS). The range for each component is 0-100 and a higher score means a better outcome.
  units on a scale | 49.0 (10.82) | 48.9 (10.31) | 48.9 (10.54)
Thermal Pain Threshold [Mean (Standard Deviation); unit: degrees Celsius] — Temperature values, measured in degrees Celsius, from 4 examiner-applied contact heat stimuli are averaged to measure the experimental thermal pain threshold (temperature at which pain is first perceived). The range was 32-50 degrees Celsius and a higher value means a better outcome.
  degrees Celsius | 41.3 (3.46) | 41.4 (3.55) | 41.3 (3.49)
Thermal Pain Tolerance [Mean (Standard Deviation); unit: degrees Celsius] — Temperature values, measured in degrees Celsius, from 4 examiner-applied contact heat stimuli are averaged to measure the experimental thermal pain tolerance (temperature at which pain can no longer be tolerated). The range was 32-50 degrees Celsius and a higher value means a better outcome.
  degrees Celsius | 45.5 (3.17) | 45.5 (3.22) | 45.5 (3.19)
Pressure Pain Threshold at Temporalis Muscle [Mean (Standard Deviation); unit: kPa] — Pressure values, measured in kiloPascals (kPa), from up to 5 experimental pressure stimuli, bilaterally applied to the area of temporalis muscle, are averaged to obtain a single pressure pain threshold value per anatomical site. The range is 0-500 kPa and a higher value means a better outcome.
  kPa | 114 (62.0) | 102 (52.9) | 108 (57.8)
Pressure Pain Threshold at Masseter Muscle [Mean (Standard Deviation); unit: kPa] — Pressure values, measured in kiloPascals (kPa), from up to 5 experimental pressure stimuli, bilaterally applied to the area of masseter muscle, are averaged to obtain a single pressure pain threshold value per anatomical site. The range is 0-500 kPa and a higher value means a better outcome.
  kPa | 106 (56.4) | 95 (53.9) | 101 (55.3)
Pressure Pain Threshold at Temporomandibular Joint [Mean (Standard Deviation); unit: kPa] — Pressure values, measured in kiloPascals (kPa), from up to 5 experimental pressure stimuli, bilaterally applied to the area of temporomandibular joint, are averaged to obtain a single pressure pain threshold value per anatomical site. The range is 0-500 kPa and a higher value means a better outcome.
  kPa | 99 (53.4) | 91 (51.8) | 95 (52.6)
Pressure Pain Threshold at Trapezius Muscle [Mean (Standard Deviation); unit: kPa] — Pressure values, measured in kiloPascals (kPa), from up to 5 experimental pressure stimuli, bilaterally applied to the area of trapezius muscle, are averaged to obtain a single pressure pain threshold value per anatomical site. The range is 0-500 kPa and a higher value means a better outcome.
  kPa | 208 (108.0) | 194 (114.2) | 201 (111.1)
Pressure Pain Threshold at Lateral Epicondyle [Mean (Standard Deviation); unit: kPa] — Pressure values, measured in kiloPascals (kPa), from up to 5 experimental pressure stimuli, bilaterally applied to the area of lateral epicondyle, are averaged to obtain a single pressure pain threshold value per anatomical site. The range is 0-500 kPa and a higher value means a better outcome.
  kPa | 213 (100.3) | 213 (111.1) | 213 (105.6)
Pain-free Jaw Opening [Mean (Standard Deviation); unit: mm] — Measured at TMD exam. A higher value means a better outcome.
  mm | 30.0 (10.79) | 29.6 (11.58) | 29.8 (11.16)
Maximum Unassisted Jaw Opening [Mean (Standard Deviation); unit: mm] — Measured at TMD exam. A higher value means a better outcome.
  mm | 43.9 (8.44) | 44.5 (10.08) | 44.2 (9.27)
Maximum Assisted Jaw Opening [Mean (Standard Deviation); unit: mm] — Measured at TMD exam. A higher value means a better outcome.
  mm | 47.6 (8.92) | 48.9 (9.39) | 48.2 (9.16)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mm Hg] — Average of 3 repeated measures taken with a 2-minute interval.
  mm Hg | 121.8 (12.65) | 122.0 (15.19) | 121.9 (13.93)
Diastolic Blood pressure [Mean (Standard Deviation); unit: mm Hg] — Average of 3 repeated measures taken with a 2-minute interval.
  mm Hg | 72.6 (9.73) | 72.3 (10.84) | 72.5 (10.27)
Heart Rate [Mean (Standard Deviation); unit: beats per minute] — Average of 3 repeated measures taken with a 2-minute interval.
  beats per minute | 74.0 (11.72) | 73.3 (11.70) | 73.7 (11.68)

OUTCOME MEASURES:

1. Primary Outcome: Change in the Weekly Mean Pain Index After 9 Weeks of Treatment
Description: Weekly mean pain index computed as the arithmetic mean of daily pain index values during the week prior to randomization and prior to each study visit. Daily pain index is computed as pain intensity (0-100 numeric rating scale where 0 = "no pain" and 100 = "the most intense pain imaginable") multiplied by pain duration (0-100 percentage scale where percent = "percent of waking day you had facial pain") as reported in the Daily Symptom Diary and divided by 100. The pain index range is from 0 to 100. A higher score means a worse outcome.
Time Frame: Visit 1 (study day 0) and Visit 4 (study day 63 +/-7)
Population: All participants who received at least one dose of study medication and provided at least one post-baseline outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Propranolol ER | Placebo
Number analyzed (Participants) | 100 | 99
units on a scale | -13.9 [-17.4 to -10.5] | -12.1 [-15.5 to -8.7]
Statistical Analysis 1: Comparison: Propranolol ER vs Placebo; Test type: Superiority; p = 0.414, Mixed Models Analysis — P-value is not adjusted for multiple comparisons and the a priori threshold for statistical significance is 0.05; Covariates for site, baseline value, sex, race, treatment, visit, a treatment*visit interaction, and an unstructured covariance structure; LSM Difference (Final Values) = -1.8, 95% CI 2-sided [-6.2 to 2.6]

2. Secondary Outcome: Change in the Weekly Mean Pain Intensity After 9 Weeks of Treatment
Description: Weekly mean pain intensity computed as the arithmetic mean of daily pain intensity values during the week prior to randomization and prior to each study visit. Daily pain intensity is measured on 0-100 numeric rating scale where 0 = "no pain" and 100 = "the most intense pain imaginable") as reported in the Daily Symptom Diary. A higher score means a worse outcome.
Time Frame: Visit 1 (study day 0) and Visit 4 (study day 63 +/-7)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Propranolol ER | Placebo
Number analyzed (Participants) | 100 | 99
units on a scale | -17.1 [-21.1 to -13.1] | -13.6 [-17.6 to -9.7]

3. Secondary Outcome: Change in the Weekly Mean Pain Duration After 9 Weeks of Treatment
Description: Weekly mean pain duration computed as the arithmetic mean of daily pain duration values during the week prior to randomization and prior to each study visit. Daily pain duration is measured on 0-100 percentage scale where percent = "percent of waking day you had facial pain" as reported in the Daily Symptom Diary. A higher score means a worse outcome.
Time Frame: Visit 1 (study day 0) and Visit 4 (study day 63 +/-7)
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Propranolol ER | Placebo
Number analyzed (Participants) | 100 | 99
units on a scale | -17.9 [-22.8 to -13.0] | -16.6 [-21.3 to -11.7]

4. Secondary Outcome: Change in the SF-McGill Pain Questionnaire Affective Component After 9 Weeks of Treatment
Description: The SF-McGill Pain Questionnaire contains 4 affective descriptors rated on a 0-3 scale where 0 = "none," 1 = "mild," 2 = "moderate," and 3 = "severe." The item scores are summed to yield a total score ranging from 0 to 12. A higher score means a worse outcome.
Time Frame: Visit 1 (study day 0) and Visit 4 (study day 63 +/-7)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Propranolol ER | Placebo
Number analyzed (Participants) | 100 | 99
score on a scale | -2.9 [-3.7 to -2.0] | -3.1 [-3.9 to -2.2]

5. Secondary Outcome: Change in the SF-McGill Pain Questionnaire Sensory Component After 9 Weeks of Treatment
Description: The SF-McGill Pain Questionnaire contains 11 sensory descriptors rated on a 0-3 scale where 0 = "none," 1 = "mild," 2 = "moderate," and 3 = "severe." The item scores are summed to yield a total score ranging from 0 to 33. A higher score means a worse outcome.
Time Frame: Visit 1 (study day 0) and Visit 4 (study day 63 +/-7)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Propranolol ER | Placebo
Number analyzed (Participants) | 100 | 99
score on a scale | -1.9 [-2.2 to -1.6] | -1.6 [-1.9 to -1.2]

6. Secondary Outcome: Change in the SF-McGill Pain Questionnaire Present Facial Pain Intensity After 9 Weeks of Treatment
Description: Self-reported present intensity of facial pain at the moment of assessment scored on a descriptive scale where 1 = "no pain' and 6 = "excruciating pain." A higher score means worse outcome.
Time Frame: Visit 1 (study day 0) and Visit 4 (study day 63 +/-7)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Propranolol ER | Placebo
Number analyzed (Participants) | 100 | 99
units on a scale | -0.9 [-1.1 to -0.7] | -0.7 [-0.9 to -0.5]

7. Secondary Outcome: Change in the SF-McGill Pain Questionnaire Weekly Average Facial Pain Intensity After 9 Weeks of Treatment
Description: Self-reported average facial pain intensity for the last week scored on 0-100 numerical rating scale where 0 = "no pain" and 100 = "the most intense pain imaginable". A higher score means a worse outcome.
Time Frame: Visit 1 (study day 0) and Visit 4 (study day 63 +/-7)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Propranolol ER | Placebo
Number analyzed (Participants) | 100 | 99
units on a scale | -18.2 [-22.6 to -13.8] | -15.8 [-20.1 to -11.5]

8. Secondary Outcome: Change in the SF-McGill Pain Questionnaire Weekly Average Facial Pain Duration After 9 Weeks of Treatment
Description: Self-reported average facial pain duration for the last week scored on 0-100 percentage scale where percent = "percent of waking day you had facial pain". A higher score means a worse outcome.
Time Frame: Visit 1 (study day 0) and Visit 4 (study day 63 +/-7)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Propranolol ER | Placebo
Number analyzed (Participants) | 100 | 99
units on a scale | -23.6 [-29.5 to -17.8] | -21.6 [-27.3 to -16.0]

9. Secondary Outcome: Change in the SF-McGill Pain Questionnaire Weekly Fatigue After 9 Weeks of Treatment
Description: Self-reported average fatigue for the last week scored on 0-100 numerical rating scale where 0 = "no fatigue" and 100 = "the greatest imaginable." A higher score means a worse outcome.
Time Frame: Visit 1 (study day 0) and Visit 4 (study day 63 +/-7)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Propranolol ER | Placebo
Number analyzed (Participants) | 100 | 99
units on a scale | -12.0 [-17.7 to -6.3] | -11.4 [-16.9 to -5.8]

10. Secondary Outcome: Number of Participants Stratified Per Graded Chronic Pain Scale (GCPS) Grade After 9 Weeks of Treatment
Description: Individuals were classified into 6 chronic pain grades: 0 = no pain; I = low pain intensity and low pain-related disability; IIa = high pain intensity and low pain-related disability; IIb = high pain intensity and high activity interference; III = moderate pain-related disability; and IV = severe pain-related disability. For analyses, this variable was dichotomized: grades 0-IIa were combined in one category and all higher grades in another. A higher grade means a worse outcome.
Time Frame: Visit 4 (study day 63 +/-7)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Propranolol ER | Placebo
Number analyzed (Participants) | 87 | 87
Participants
  GCPS Grades 0-IIa | 75 | 69
  GCPS Grades IIb-IV | 12 | 18

11. Secondary Outcome: Change in the Jaw Functional Limitation Scale (JFLS) Global Score After 9 Weeks of Treatment
Description: The JFLS contains 20 items that measure limitations across mastication, vertical jaw mobility, and verbal/emotional expression rated on a 0-10 scale where 0 = "no limitation" and 10 = "severe limitation." The Global Score is computed as the mean response for all items and ranges from 0 to 10. A higher score means a worse outcome.
Time Frame: Visit 1 (study day 0) and Visit 4 (study day 63 +/-7)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Propranolol ER | Placebo
Number analyzed (Participants) | 100 | 99
score on a scale | -1.1 [-1.4 to -0.8] | -0.8 [-1.1 to -0.6]

12. Secondary Outcome: Change in the Headache Impact Test (HIT-6) Global Score After 9 Weeks of Treatment
Description: The HIT-6 contains 6 items and assesses headache-related disability by the frequency of daily activity limitations ranging from "never" to "always." The 6 item scores are summed to yield a global score ranging from 36 to 78. A higher score means a worse outcome.
Time Frame: Visit 1 (study day 0) and Visit 4 (study day 63 +/-7)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Propranolol ER | Placebo
Number analyzed (Participants) | 100 | 99
score on a scale | -5.1 [-6.6 to -3.6] | -3.1 [-4.6 to -1.7]

13. Secondary Outcome: Change in the Pittsburgh Sleep Quality Index (PSQI) Global Score After 9 Weeks of Treatment
Description: The PSQI has 19 items grouped into 7 component scores, each weighted equally on a 0-3 scale, The 7 component scores are summed to yield a global PSQI score, which has a range of 0-21. A higher score means a worse outcome.
Time Frame: Visit 1 (study day 0) and Visit 4 (study day 63 +/-7)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Propranolol ER | Placebo
Number analyzed (Participants) | 100 | 99
score on a scale | -0.7 [-1.3 to 0.0] | -1.0 [-1.6 to -0.4]

14. Secondary Outcome: Number of Participants Stratified Per Dichotomized Score From the Patient Global Impression of Change (PGIC) Scale After 9 Weeks of Treatment
Description: The PGIC scale assesses patient overall change in the severity of illness following treatment. Participants rate how they feel now compared with how they felt before receiving study drug on a 7-point scale where 0 = "No change or condition has got worse" and 6 = "A great deal better." A higher score means a better outcome. For analyses, this variable was dichotomized: scores from 0 to 3 were combined in one category of "No" (no significant improvement) and scores from 4 to 6 were combined in another category of "Yes" (significant improvement with the study treatment).
Time Frame: Visit 4 (study day 63 +/-7)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Propranolol ER | Placebo
Number analyzed (Participants) | 87 | 87
Participants
  No | 46 | 60
  Yes | 41 | 27

15. Secondary Outcome: Change in the Perceived Stress Scale (PSS) Global Score After 9 Weeks of Treatment
Description: The PSS assesses the frequency of 14 sources of stress on a scale from 0 = "never" to 4 = "very often." The item scores are summed to yield a global score ranging from 0 to 56. A higher score means a worse outcome.
Time Frame: Visit 1 (study day 0) and Visit 4 (study day 63 +/-7)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Propranolol ER | Placebo
Number analyzed (Participants) | 100 | 99
score on a scale | -2.6 [-4.1 to -1.1] | -1.9 [-3.4 to -0.5]

16. Secondary Outcome: Change in the Hospital Anxiety and Depression Scale (HADS) Depression Score After 9 Weeks of Treatment
Description: The HADS is a 14-item assessment of anxiety (7 items) and depression (7 items) using the relative frequency of symptoms over the past week, rated on a 4-point scale ranging from 0 = "not at all" to 3 = "very often indeed". Responses are summed to provide separate scores for anxiety and depression with a range from 0 to 21. A higher score means a worse outcome.
Time Frame: Visit 1 (study day 0) and Visit 4 (study day 63 +/-7)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Propranolol ER | Placebo
Number analyzed (Participants) | 100 | 99
score on a scale | -1.0 [-1.6 to -0.4] | -0.6 [-1.1 to 0.0]

17. Secondary Outcome: Change in the Hospital Anxiety and Depression Scale (HADS) Anxiety Score After 9 Weeks of Treatment
Description: as for outcome 16
Time Frame: Visit 1 (study day 0) and Visit 4 (study day 63 +/-7)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Propranolol ER | Placebo
Number analyzed (Participants) | 100 | 99
score on a scale | -1.3 [-2.0 to -0.7] | -0.7 [-1.3 to -0.1]

18. Secondary Outcome: Change in the Symptom Checklist 90-Revised (SCL-90R) Somatization Scale Score After 9 Weeks of Treatment
Description: The SCL-90R Somatization Scale is a 12-item assessment of somatic symptom distress over the past 7 days rated from 0 = "not at all" to 4 = "extremely." The scale score is computed as the mean for all items. The score range is from 0 to 4. A higher score means a worse outcome.
Time Frame: Visit 1 (study day 0) and Visit 4 (study day 63 +/-7)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Propranolol ER | Placebo
Number analyzed (Participants) | 100 | 99
score on a scale | -0.2 [-0.3 to -0.1] | -0.2 [-0.3 to -0.1]

19. Secondary Outcome: Change in the SF-12 Health Survey v2 (SF-12v2) Physical Component Summary (PCS) After 9 Weeks of Treatment
Description: The SF-12v2 contains 7 questions assessing 8 domains of functioning and well-being rated from: "excellent" to "poor" (for general health); "yes, limited a lot" to "no, not limited at all" (for functional level); and "all of the time" to "none of the time" (for emotional state). These 8 domains can be further summarized into a physical component summary (PCS) and a mental component summary (MCS). summary (MCS). The range for each component is 0-100 and a higher score means a better outcome.
Time Frame: Visit 1 (study day 0) and Visit 4 (study day 63 +/-7)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Propranolol ER | Placebo
Number analyzed (Participants) | 100 | 99
score on a scale | 1.2 [-0.3 to 2.6] | 0.3 [-1.2 to 1.7]

20. Secondary Outcome: Change in the SF-12 Health Survey v2 (SF-12v2) Mental Component Summary (MCS) After 9 Weeks of Treatment
Description: The SF-12v2 contains 7 questions assessing 8 domains of functioning and well-being rated from: "excellent" to "poor" (for general health); "yes, limited a lot" to "no, not limited at all" (for functional level); and "all of the time" to "none of the time" (for emotional state). These 8 domains can be further summarized into a physical component summary (PCS) and a mental component summary (MCS). The range for each component is 0-100 and a higher score means a better outcome.
Time Frame: Visit 1 (study day 0) and Visit 4 (study day 63 +/-7)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Propranolol ER | Placebo
Number analyzed (Participants) | 100 | 99
score on a scale | 3.6 [1.6 to 5.6] | 2.8 [0.9 to 4.8]

21. Secondary Outcome: Change in Thermal Pain Threshold After 9 Weeks of Treatment
Description: Temperature values, measured in degrees Celsius, from 4 examiner-applied contact heat stimuli will be averaged to measure the experimental thermal pain threshold (temperature at which pain is first perceived). The range was 32-50 degrees Celsius and a higher value means a better outcome.
Time Frame: Visit 1 (study day 0) and Visit 4 (study day 63 +/-7)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: degrees Celsius
Arm/Group | Propranolol ER | Placebo
Number analyzed (Participants) | 100 | 99
degrees Celsius | 1.3 [0.7 to 1.9] | 0.5 [-0.1 to 1.1]

22. Secondary Outcome: Change in Thermal Pain Tolerance After 9 Weeks of Treatment
Description: Temperature values, measured in degrees Celsius, from 4 examiner-applied contact heat stimuli will be averaged to measure the experimental thermal pain tolerance (temperature at which pain can no longer be tolerated). The range was 32-50 degrees Celsius and a higher value means a better outcome.
Time Frame: Visit 1 (study day 0) and Visit 4 (study day 63 +/-7)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: degrees Celsius
Arm/Group | Propranolol ER | Placebo
Number analyzed (Participants) | 100 | 99
degrees Celsius | 0.5 [0.2 to 0.9] | 0.4 [0.0 to 0.8]

23. Secondary Outcome: Change in Pressure Pain Threshold at Temporalis Muscle After 9 Weeks of Treatment
Description: Pressure values, measured in kilopascals (kPa), from up to 5 experimental pressure stimuli, bilaterally applied to the area of temporalis muscle, are averaged to obtain a single pressure pain threshold value per anatomical site. The range is 0-500 kPa and a higher value means a better outcome.
Time Frame: Visit 1 (study day 0) and Visit 4 (study day 63 +/-7)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: kPa
Arm/Group | Propranolol ER | Placebo
Number analyzed (Participants) | 100 | 99
kPa | 41.8 [29.0 to 54.7] | 38.4 [26.2 to 50.6]

24. Secondary Outcome: Change in Pressure Pain Threshold at Masseter Muscle After 9 Weeks of Treatment
Description: Pressure values, measured in kilopascals, from up to 5 experimental pressure stimuli, bilaterally applied to the area of masseter muscle, will be averaged to obtain a single pressure pain threshold value per anatomical site.
Time Frame: Visit 1 (study day 0) and Visit 4 (study day 63 +/- 7)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: kPa
Arm/Group | Propranolol ER | Placebo
Number analyzed (Participants) | 100 | 99
kPa | 38.3 [26.6 to 50.0] | 29.3 [18.2 to 40.4]

25. Secondary Outcome: Change in Pressure Pain Threshold at Temporomandibular Joint After 9 Weeks of Treatment
Description: Pressure values, measured in kilopascals, from up to 5 experimental pressure stimuli, bilaterally applied to the area of temporomandibular joint, will be averaged to obtain a single pressure pain threshold value per anatomical site.
Time Frame: Visit 1 (study day 0) and Visit 4 (study day 63 +/-7)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: kPa
Arm/Group | Propranolol ER | Placebo
Number analyzed (Participants) | 100 | 99
kPa | 36.8 [26.6 to 47.0] | 25.3 [15.4 to 35.1]

26. Secondary Outcome: Change in Pressure Pain Threshold at Trapezius Muscle After 9 Weeks of Treatment
Description: Pressure values, measured in kilopascals, from up to 5 experimental pressure stimuli, bilaterally applied to the area of trapezius muscle, will be averaged to obtain a single pressure pain threshold value per anatomical site.
Time Frame: Visit 1 (study day 0) and Visit 4 (study day 63 +/-7)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: kPa
Arm/Group | Propranolol ER | Placebo
Number analyzed (Participants) | 100 | 99
kPa | 64.1 [41.1 to 87.2] | 63.3 [41.1 to 85.5]

27. Secondary Outcome: Change in Pressure Pain Threshold at Lateral Epicondyle After 9 Weeks of Treatment
Description: Pressure values, measured in kilopascals, from up to 5 experimental pressure stimuli, bilaterally applied to the area of lateral epicondyle, will be averaged to obtain a single pressure pain threshold value per anatomical site.
Time Frame: Visit 1 (study day 0) and Visit 4 (study day 63 +/-7)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: kPa
Arm/Group | Propranolol ER | Placebo
Number analyzed (Participants) | 100 | 99
kPa | 41.4 [22.2 to 60.7] | 22.7 [4.0 to 41.5]

28. Secondary Outcome: Change in Pain-free Jaw Opening After 9 Weeks of Treatment
Description: Measured at TMD exam. A higher value means a better outcome.
Time Frame: Visit 1 (study day 0) and Visit 4 (study day 63 +/-7)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mm
Arm/Group | Propranolol ER | Placebo
Number analyzed (Participants) | 100 | 99
mm | 4.5 [1.3 to 7.7] | 1.4 [-1.6 to 4.4]

29. Secondary Outcome: Change in Maximum Unassisted Jaw Opening After 9 Weeks of Treatment
Description: Measured at TMD exam. A higher value means a better outcome.
Time Frame: Visit 1 (study day 0) and Visit 4 (study day 63 +/-7)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mm
Arm/Group | Propranolol ER | Placebo
Number analyzed (Participants) | 100 | 99
mm | -0.9 [-3.2 to 1.4] | -1.2 [-3.4 to 0.9]

30. Secondary Outcome: Change in Maximum Assisted Jaw Opening After 9 Weeks of Treatment
Description: Measured at TMD exam. A higher value means a better outcome.
Time Frame: Visit 1 (study day 0) and Visit 4 (study day 63 +/-7)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mm
Arm/Group | Propranolol ER | Placebo
Number analyzed (Participants) | 100 | 99
mm | -0.3 [-2.3 to 1.8] | -0.8 [-2.7 to 1.1]

31. Secondary Outcome: Change in Systolic Blood Pressure After 9 Weeks of Treatment
Description: Average of 3 repeated measures taken with a 2-minute interval.
Time Frame: Visit 1 (study day 0) and Visit 4 (study day 63 +/-7)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mm Hg
Arm/Group | Propranolol ER | Placebo
Number analyzed (Participants) | 100 | 99
mm Hg | -3.6 [-5.7 to -1.5] | 1.3 [-0.8 to 3.4]

32. Secondary Outcome: Change in Diastolic Blood Pressure After 9 Weeks of Treatment
Description: Average of 3 repeated measures taken with a 2-minute interval.
Time Frame: Visit 1 (study day 0) and Visit 4 (study day 63 +/-7)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mm Hg
Arm/Group | Propranolol ER | Placebo
Number analyzed (Participants) | 100 | 99
mm Hg | -3.3 [-4.9 to -1.8] | 1.0 [-0.5 to 2.5]

33. Secondary Outcome: Change in Heart Rate After 9 Weeks of Treatment
Description: Average of 3 repeated measures taken with a 2-minute interval.
Time Frame: Visit 1 (study day 0) and Visit 4 (study day 63 +/-7)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: beats per minute
Arm/Group | Propranolol ER | Placebo
Number analyzed (Participants) | 100 | 99
beats per minute | -3.9 [-5.8 to -2.0] | 1.5 [-0.4 to 3.3]

34. Other Pre Specified Outcome: Change in the Weekly Mean Pain Index After 9 Weeks of Treatment Stratified Per Number of COMT LPS Haplotypes
Description: Weekly mean pain index computed as the arithmetic mean of daily pain index values during the week prior to randomization and prior to each study visit. Daily pain index is computed as pain intensity (0-100 numeric rating scale where 0 = "no pain" and 100 = "the most intense pain imaginable") multiplied by pain duration (0-100 percentage scale where percent = "percent of waking day you had facial pain") as reported in the Daily Symptom Diary, divided by 100. The pain index range is from 0 to 100. A higher score means a worse outcome. The pain index was stratified per number of catechol-O-methyltransferase (COMT) Low Pain Sensitive (LPS) haplotypes.
Time Frame: Visit 1 (study day 0) and Visit 4 (study day 63 +/-7)
Population: All participants who received at least one dose of study medication, provided at least one post-baseline outcome measure, and had genotyping data for COMT haplotypes.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Propranolol ER | Placebo
Number analyzed (Participants) | 82 | 85
units on a scale
  0 LPS haplotypes: number analyzed (Participants) | 31 | 36
  0 LPS haplotypes | -14.2 [-19.3 to -9.2] | -12.3 [-17.3 to -7.4]
  1 LPS haplotype: number analyzed (Participants) | 37 | 43
  1 LPS haplotype | -12.2 [-17.3 to -7.0] | -13.2 [-17.9 to -8.5]
  2 LPS haplotypes: number analyzed (Participants) | 14 | 6
  2 LPS haplotypes | -15.2 [-23.3 to -7.0] | -2.5 [-13.6 to 8.7]

35. Other Pre Specified Outcome: Change in the Weekly Mean Pain Index After 9 Weeks of Treatment Stratified Per Number of COMT Valine Alleles at rs4680
Description: Weekly mean pain index computed as the arithmetic mean of daily pain index values during the week prior to randomization and prior to each study visit. Daily pain index is computed as pain intensity (0-100 numeric rating scale where 0 = "no pain" and 100 = "the most intense pain imaginable") multiplied by pain duration (0-100 percentage scale where percent = "percent of waking day you had facial pain") as reported in the Daily Symptom Diary, divided by 100. The pain index range is from 0 to 100. A higher score means a worse outcome. The pain index was stratified per number of catechol-O-methyltransferase (COMT) valine alleles at single nucleotide polymorphism (SNP) rs4680.
Time Frame: Visit 1 (study day 0) and Visit 4 (study day 63 +/-7)
Population: All participants who received at least one dose of study medication, provided at least one post-baseline outcome measure, and had genotyping data for COMT rs4680.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Propranolol ER | Placebo
Number analyzed (Participants) | 83 | 85
units on a scale
  0 valine alleles: number analyzed (Participants) | 19 | 16
  0 valine alleles | -14.2 [-20.9 to -7.6] | -13.9 [-21.5 to -6.3]
  1 valine allele: number analyzed (Participants) | 34 | 46
  1 valine allele | -13.9 [-19.2 to -8.6] | -13.1 [-17.6 to -8.6]
  2 valine alleles: number analyzed (Participants) | 30 | 23
  2 valine alleles | -14.3 [-19.7 to -9.0] | -9.7 [-15.8 to -3.6]

ADVERSE EVENTS:
Time Frame: From obtaining informed consent until 7 (for nonserious AEs) or 30 days (for SAEs) after the last day of study participation.
Description: 8 AEs commonly reported with use of propranolol were solicited by a questionnaire administered at each study visit. All the rest of the AEs were solicited through the open-question inquiries at each study visit. Data are reported for AEs that occurred in the safety sample which includes all randomized participants who received at least one dose of study medication. Participants are analyzed according to the medication they actually received, regardless of their randomized assignment.
Arm/Group | Propranolol ER | Placebo
All-Cause Mortality (participants affected / at risk) | 1/100 | 0/100
Serious Adverse Events (participants affected / at risk) | 4/100 | 1/100
Other Adverse Events (participants affected / at risk) | 86/100 | 75/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Propranolol ER (N=100) | Placebo (N=100)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0) — Occurred in a participant with metastatic breast cancer
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0) — Occurred in a participant with metastatic breast cancer
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Alcohol abuse (Psychiatric disorders) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Propranolol ER (N=100) | Placebo (N=100)
Diarrhoea (Gastrointestinal disorders) | 20 (23) | 18 (22)
Nausea (Gastrointestinal disorders) | 19 (20) | 9 (9)
Constipation (Gastrointestinal disorders) | 10 (13) | 10 (10)
Vomiting (Gastrointestinal disorders) | 5 (5) | 3 (3)
Fatigue (General disorders) | 32 (38) | 21 (24)
Dizziness (Nervous system disorders) | 25 (31) | 9 (10)
Paraesthesia (Nervous system disorders) | 7 (8) | 13 (14)
Hypoaestesia (Nervous system disorders) | 6 (7) | 8 (8)
Headache (Nervous system disorders) | 5 (5) | 1 (1)
Migraine (Nervous system disorders) | 5 (7) | 0 (0)
Nasopharyngitis (Infections and infestations) | 13 (15) | 12 (12)
Upper respiratory tract infection (Infections and infestations) | 7 (8) | 7 (7)
Insomnia (Psychiatric disorders) | 16 (20) | 12 (13)
Depression (Psychiatric disorders) | 10 (12) | 10 (11)
Sleep disorder (Psychiatric disorders) | 6 (8) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 6 (6)
Injury (Injury, poisoning and procedural complications) | 10 (12) | 9 (10)
Vertigo (Ear and labyrinth disorders) | 6 (7) | 7 (7)
Skin and subcutaneos tissue disorders (Skin and subcutaneous tissue disorders) | 6 (8) | 8 (8)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 7 (11) | 3 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-02-12): https://cdn.clinicaltrials.gov/large-docs/83/NCT02437383/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-21): https://cdn.clinicaltrials.gov/large-docs/83/NCT02437383/SAP_001.pdf